CLINICAL TRIAL: NCT00522444
Title: Nebulized Magnesium Sulfate Compared to Saline in Addition to Albuterol and Ipratropium Treatments in Moderate to Severe Pediatric Asthmatic Patients: A Randomized Controlled Clinical Trial
Brief Title: Nebulized Magnesium Sulfate in Pediatric Asthma
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-0431
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- nebulized magnesium sulfate (Experimental): 6.3% solution of magnesium heptahydrate, which is equivalent to 3.18% anhydrous magnesium sulfate
  Interventions: Drug: Nebulized Magnesium Sulfate
- normal saline nebulization (Placebo Comparator): standard of care
  Interventions: Other: Nebulized normal saline

INTERVENTIONS:
Drug: Nebulized Magnesium Sulfate — 6.3% solution of magnesium heptahydrate, which is equivalent to 3.18% anhydrous magnesium sulfate
  Other Names: magnesium heptahydrate
  Arms: nebulized magnesium sulfate
Other: Nebulized normal saline — standard of care
  Arms: normal saline nebulization

SUMMARY:
Nebulized Magnesium Sulfate has been shown to be of benefit in adults with acute asthma exacerbations, though limited work has been done in the pediatric population. Current therapeutic questions include the effect of more than one dose of nebulized magnesium, the possibility of a sustained effect (greater than 20 minutes) after a treatment, the potential benefit in children younger than 5 years of age, and the use of an asthma score to re-assess patients after treatment with this medication. The purpose of this double-blind randomized placebo-controlled clinical trial is the evaluate the effect of multiple doses of nebulized magnesium sulfate versus saline in addition to standard asthma therapy on clinical asthma score and FEV1 in children 7 to 18 years of age with a moderate to severe acute asthma exacerbation. Our hypothesis is that nebulized magnesium sulfate, when added to traditional bronchodilator therapy, will improve acute asthma exacerbations more rapidly than standard therapy alone. The primary outcomes are asthma score and FEV1 values obtained after two nebulized magnesium sulfate compared to placebo treatments. This therapy will be supplemental to standard therapy of albuterol and ipratropium nebulized treatments and systemic corticosteroids. The secondary outcome is patient disposition (discharge home or hospitalization). Patients with known asthma will be approached for enrollment and informed consent obtained if the asthma score after the first albuterol treatment is "2" or greater. One hundred-seventy patients will be enrolled and randomized to either the treatment group or the placebo group. The change from baseline in asthma scores and FEV1 values will be compared among the control and treatment groups to assess for any benefit of the addition of nebulized magnesium sulfate to the treatment regimen.

DETAILED DESCRIPTION:
Acute asthma exacerbations continue to be a growing heath care dilemma, even as increased efforts are made in preventing such exacerbations. The standard of care for such exacerbations typically involves inhaled beta-agonist therapy and oral steroids. Patients who are refractory to these treatments may require intravenous access for the purposes of delivering additional medications, including magnesium sulfate. Intravenous magnesium sulfate has been shown to be beneficial in moderate and severe acute asthma exacerbations in adults and children, and new research indicates a trend toward benefits from nebulized magnesium sulfate, even in those with a mild exacerbation of asthma. Delivery of magnesium sulfate via the inhalation route is less invasive than the intravenous route, which is preferable in the pediatric population. The possible short-term benefits of the nebulized form of magnesium sulfate include decreased ED length of stay and prevention of admission to the intensive care unit if the patient must be hospitalized for further treatments. The specific aim of this study is to evaluate the effect of the addition of nebulized magnesium sulfate to our standard emergency department therapy by comparing the change from baseline of asthma scores and FEV1 (forced expiratory volume in 1 second) in children with acute asthma exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Patients ages 7-18 years old
* Parental report of previous history of asthma or wheezing episode documented by physician at least 3 months prior to enrollment
* Acute Asthma exacerbation as defined by attending physician and asthma score (PASS) of greater than or equal to 2 after initial albuterol treatment

Exclusion Criteria:

* Temperature in triage of greater than or equal to 39 degrees Celsius
* Systemic corticosteroids in past 72 hours
* Medical history significant for cardiac, renal, or malignant disease, or bronchopulmonary dysplasia or cystic fibrosis
* Patients whose care is initiated in the trauma bay due to need for rapid stabilization or any patient deemed too ill to participate by the attending ED physician
* Altered Mental Status (Glasgow Coma Score of < 15)
* Asthma Score (PASS) of > 6, and in conjunction with FEV1 < 45% predicted
* Oxygen saturation < 90% while on 6L of 100% oxygen via face mask
* Respiratory distress occurring after FEV1 attempt in conjunction with any increase in asthma score (PASS) from previous score
* Enrollment in any other research study in the previous 30 days
* Previous enrollment in this RCT
* Initial administration of continuously nebulized albuterol or dose of IV Magnesium Sulfate in the ED

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change is PASS Asthma Score | through emergency admission, an average of less than 1 day
  The primary outcome event for the assessment of efficacy in all patients is the change in PASS asthma score from Time Zero to Times One and Two.

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Johnson, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati